CLINICAL TRIAL: NCT06629129
Title: Optic Nerve Head Perfusion Following Treatment with Latanoprost 0.005% in Primary Open Angle Glaucoma: an Optical Coherence Tomography Angiography Study
Brief Title: Effect of Latanoprost on Optic Nerve Perfusion
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #454/25-June-2024
Record Dates: First submitted 2024-09-28; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Treatment Outcome
Keywords: Open angle glaucoma; OCTA; RNFL
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Latanoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- EFFECT OF ANTI GLAUCOMA LATANOPROST 0.005 ON OPTIC NERVE PERFUSION (Other): EFFECT OF ANTI GLAUCOMA PROSTAGLANDIN 0.005 ON OPTIC NERVE PERFUSION
  Interventions: Drug: Latanoprost (0.005%)

INTERVENTIONS:
Drug: Latanoprost (0.005%) — MEAN OCULAR PERFUSION PRESSURE WAS MEASURED AND CORRELATED TO THE IOP AND OPTIC NERVE PERFUSION IN RESPONSE TO LATANOPROST TREATMENT

SUMMARY:
46 eyes of 23 patients have been treated with topical Latanoprost 0.005 %. visual field was performed on all eyes. NFLT was measured using OCT. Radial peripapillary capillary (RPC) vascular density was measured using OCTA . mean ocular perfusion pressure (MOPP), and RPC vascular density were measured before and after treatment BY 2-3 MONTHS

DETAILED DESCRIPTION:
All patients had bilateral primary open angle glaucoma diagnosed by increased IOP, visual field changes, and defective nerve fiber layer thickness (NFLT) on OCT examination.

All patients treated with topical Latanoprost 0.005% (XalatanTM, 2.5 ml eye drops, Pfizer) Inclusion criteria: age > 20 years, newly diagnosed patients with POAG. The exclusion criteria included optic nerve lesions other than glaucomatous changes, All patients completed their ophthalmic examination to detect BCVA, cycloplegic refraction, and anterior segment examination , IOP measuring by applanation tonometer, and indirect ophthalmoscope fundus examination.

Visual field testing. The thickness of NFL around the disc was evaluated using spectral domain optical coherence tomography (OCT) Optovue octa was used to quantify the density of the radial peripapillary capillary (RPC) vessels. This study employed software to quantify the capillary (microvasculature) density in both the entire image and in the peripapillary region specifically the superior, nasal, inferior, and temporal quadrants.

The mean arterial blood pressure (MAP) was determined by adding the diastolic blood pressure (DBP) to one third of the difference between systolic blood pressure and the diastolic blood pressure.

All eyes were treated with topical latanoprost 0.005% (XalatanTM, 2.5 ml eye drops, Pfizer) with dose of one drop at bedtime. IOP, MOPP, NFLT, and RPC vascular density were measured before the beginning of treatment and 1 and 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

POAG with no past ocular surgery or laser retinal treatment. No previous anti-glaucoma medications

Exclusion Criteria:

* optic nerve lesions other than glaucoma

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
quantify the peri papillary capillary (microvasculature) density using OCTA | 3 months
  quantify the capillary (microvasculature) density in both the entire image and in the peripapillary region specifically the superior, nasal, inferior, and temporal quadrants

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris A, Migliardi R, Rechtman E, Cole CN, Yee AB, Garzozi HJ. Comparative analysis of the effects of dorzolamide and latanoprost on ocular hemodynamics in normal tension glaucoma patients. Eur J Ophthalmol. 2003 Jan-Feb;13(1):24-31. doi: 10.1177/112067210301300104. PMID 12635671
- [Background] Gherghel D, Hosking SL, Cunliffe IA, Armstrong RA. First-line therapy with latanoprost 0.005% results in improved ocular circulation in newly diagnosed primary open-angle glaucoma patients: a prospective, 6-month, open-label study. Eye (Lond). 2008 Mar;22(3):363-9. doi: 10.1038/sj.eye.6702639. Epub 2006 Nov 17. PMID 17115020